CLINICAL TRIAL: NCT04764968
Title: Pen-Administered Low-Dose Dasiglucagon for Prevention and Treatment of Hypoglycemia in People With Type 1 Diabetes: A Randomized, Open-Label, Two-Period Crossover Outpatient Study
Brief Title: Pen-Administered Low-Dose Dasiglucagon for Prevention and Treatment of Hypoglycemia in People With Type 1 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Steno Diabetes Center Copenhagen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 77119; H-21000002 (Other: Regional Scientific Ethics Committee); 2020-005745-16 (EudraCT Number)
Record Dates: First submitted 2021-02-16; First posted 2021-02-21 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Type 1 Diabetes; Hypoglycemia
Keywords: Type 1 Diabetes; Hypoglycemia; Dasiglucagon
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia | interventions — dasiglucagon

STUDY DESIGN:
Intervention Model Description: A Randomized, Open-Label, Two-Period, Two-Week Crossover Outpatient Study
Masking Description: Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (No Intervention): During the 'usual care' period, participants will manage episodes of manifest or impending hypoglycemia as usual, e.g. through carbohydrate consumption or manual insulin pump suspension.
- Dasiglucagon (Experimental): During the 'dasiglucagon' period, participants will use pen-administered low-dose (80 µg) dasiglucagon to treat or prevent episodes of hypoglycemia.
  Interventions: Drug: Dasiglucagon

INTERVENTIONS:
Drug: Dasiglucagon — Abdominal s.c. administration using a multi-dose reusable pen injector
  Arms: Dasiglucagon

SUMMARY:
The aim of the study is to evaluate the efficacy, safety and feasibility of outpatient-utilization of low-dose dasiglucagon administered via a multi-dose reusable pen injector in preventing and treating mild hypoglycemia in insulin pump-treated people with type 1 diabetes.

DETAILED DESCRIPTION:
A randomized, open-label, two-arm, two-week crossover study will be conducted to assess the study objectives. The study will enroll 24 participants with insulin pump-treated type 1 diabetes. Upon study enrollment, participants will complete two consecutive 2-week periods - a 'usual care' period and 'dasiglucagon' period. During the 'usual care' period, participants will manage episodes of manifest or impending hypoglycemia as usual, e.g. through carbohydrate consumption or manual insulin pump suspension. During the 'dasiglucagon' period, participants will use pen-administered low-dose dasiglucagon to treat or prevent episodes of hypoglycemia.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* T1D ≥ 2 years
* Use of insulin pump therapy (without sensor-augmented insulin suspension/adjustment functionality) ≥ 6 months
* Use of CGM (real-time or intermittently scanned) ≥ 3 months and ≥ 70% during the previous 14 days
* HbA1c ≤ 70 mmol/l (8.5%)
* Performs aerobic exercise on a regular basis (≥ 2 times per week; self-reported) and desires to exercise per American Diabetes Association guidelines (150 minutes per week) during the study.
* Use of carbohydrate counting and bolus calculator (self-reported)
* Sensor glucose level < 3.9 mmol/l on ≥ 4/14 previous days assessed by CGM data

Exclusion Criteria:

* Use of anti-diabetic medicine (other than insulin), corticosteroids or other drugs affecting glucose metabolism during the study period and within 30 days prior to study start
* Known or suspected allergies to glucagon or related products
* History of hypersensitivity or allergic reaction to dasiglucagon or any of the excipients
* Patients with pheochromocytoma or insulinoma
* Hypoglycemia unawareness
* Females of childbearing potential who are pregnant, breast-feeding or intend to become pregnant or are not using adequate contraceptive methods
* Inability to understand the individual information and to give informed consent
* Current participation in another clinical trial that, in the judgment of the investigator, will compromise the results of the study or the safety of the subject
* Concomitant medical or psychological conditions identified through review of medical history, physical examination and clinical laboratory analysis that, according to the investigator's assessment, makes the individual unsuitable for study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-04-27 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-01-28 (Actual)

PRIMARY OUTCOMES:
Difference in percentage of time in range between the two study periods | 2-week 'usual care' period and 2-week 'dasiglucagon' period
  Sensor glucose level ≥ 3.9 mmol/l and ≤ 10.0 mmol/l

SECONDARY OUTCOMES:
Difference in percentage of time in hypoglycemia between the two study periods | 2-week 'usual care' period and 2-week 'dasiglucagon' period
  Sensor glucose level < 3.9 mmol/l
Difference in percentage of time in hyperglycemia between the two study periods | 2-week 'usual care' period and 2-week 'dasiglucagon' period
  Sensor glucose level > 10 mmol/l
Difference in coefficient of variation (%) between the two study periods | 2-week 'usual care' period and 2-week 'dasiglucagon' period
Difference between successful cases (%) of hypoglycemia treatment between the two study periods | 2-week 'usual care' period and 2-week 'dasiglucagon' period
  Initial sensor glucose level ≥ 2.2 mmol/l and ≤ 3.9 mmol/l AND sensor glucose level > 3.9 mmol/l 30 minutes post-treatment
Difference in successful cases (%) of hypoglycemia treatment without subsequent hyperglycemia [sensor glucose level > 10 mmol/l during the first two hours post-treatment] between the two study periods | 2-week 'usual care' period and 2-week 'dasiglucagon' period
  Initial sensor glucose level ≥ 2.2 mmol/l and ≤ 3.9 mmol/l AND sensor glucose level > 3.9 mmol/l 30 minutes post-treatment AND sensor glucose level ≤ 10 mmol/l during the first two hours post-treatment
Difference in successful cases (%) of hypoglycemia prevention between the two study periods | 2-week 'usual care' period and 2-week 'dasiglucagon' period
  Initial sensor glucose level > 3.9 mmol/l AND sensor glucose level < 3.9 for ≤ 15 consecutive minutes during the first two hours post-treatment
Difference in time from hypoglycemia treatment to euglycemia between the two study periods | 2-week 'usual care' period and 2-week 'dasiglucagon' period
  Minutes from initial sensor glucose level ≥ 2.2 mmol/l and ≤ 3.9 mmol/l to sensor glucose level ≥ 3.9 mmol/l
Incidence rate of supplement carbohydrate administration during the first hour following dasiglucagon administration | 2-week 'dasiglucagon' period
Difference between the average daily carbohydrate intake between the two study periods | 2-week 'usual care' period and 2-week 'dasiglucagon' period
  Registered on the insulin pump
Difference between the average total daily insulin dose between the two study periods | 2-week 'usual care' period and 2-week 'dasiglucagon' period
Difference in the number and intensity of episodes with nausea, headache, stomach-ache, palpitations and injection site pain between the two study periods | 2-week 'usual care' period and 2-week 'dasiglucagon' period
  Intensity: mild/moderate/severe
Percentage of participants scoring a favorable outcome on the patient-reported outcome questionnaire | At the end-of-study visit (estimated week 6)
  Scoring likely OR very likely on a four-point Likert scale
Percentage of participants with treatment-induced or treatment-boosted anti-dasiglucagon antibodies | Measured 4 weeks after the 'dasiglucagon' period

OTHER OUTCOMES:
Number of device failures/malfunctions | 2-week 'dasiglucagon' period

CONTACTS AND LOCATIONS:
Overall Officials: Christian Laugesen, MD, Principal Investigator — Steno Diabetes Center Copenhagen
Locations (1):
- Steno Diabetes Center Copenhagen, Gentofte Municipality, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Laugesen C, Ranjan AG, Schmidt S, Norgaard K. Pen-administered low-dose dasiglucagon vs usual care for prevention and treatment of non-severe hypoglycaemia in people with type 1 diabetes during free-living conditions: a Phase II, randomised, open-label, two-period crossover trial. Diabetologia. 2023 Jul;66(7):1208-1217. doi: 10.1007/s00125-023-05909-4. Epub 2023 Apr 11. PMID 37037948